CLINICAL TRIAL: NCT01171287
Title: Effects of Right Lower Limb Orthopedic Immobilization on Braking Function : An On-the-Road Experimental Study by Healthy Volunteers
Brief Title: Effects of Right Lower Limb Orthopedic Immobilization on Braking Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); BSN Medical Inc (Industry)
Responsible Party: Principal Investigator, Francois Cabana, Doctor, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Erica 02
Record Dates: First submitted 2010-07-19; First posted 2010-07-28 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Automobile Driving With an Aircast Walker; Automobile Driving With a Walking Cast
Keywords: Automobile Driving; Fracture Fixation/instrumentation; Lower Extremity; Orthopedic Fixation Devices; Orthopedic Procedures; Reaction Time; Task Performance and Analysis; Time Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aircast Walker (Experimental): Automobile driving with an Aircast Walker applied to each participant's right lower extremity
  Interventions: Procedure: Driving with an Aircast Walker
- Walking cast (Experimental): Automobile driving with a walking cast applied to each participant's right lower extremity
  Interventions: Procedure: Driving with a walking cast
- Running shoe (Active Comparator): Automobile driving with a running shoe applied to each participant's right lower extremity
  Interventions: Procedure: Driving with a running shoe

INTERVENTIONS:
Procedure: Driving with an Aircast Walker
  Arms: Aircast Walker
Procedure: Driving with a walking cast
  Arms: Walking cast
Procedure: Driving with a running shoe
  Arms: Running shoe

SUMMARY:
Research on the implications of orthopedic injury and surgery on automobile driving ability has been limited. Only a handful of orthopedic issues have been studied to date, especially the safe postoperative resumption of driving. However, effects of orthopedic immobilizations of the lower right limb on fitness to drive are largely unknown, and the physician is left with little guidance. Only one study (Tremblay et al. 2009) have looked at the impact of wearing such devices on braking performances. The results have shown a statistically significant increase of braking times while wearing a removable Aircast walker and a walking cast in healthy subjects under simulated driving conditions. Despite this, the study have not demonstrated that driving with orthopedic immobilization is dangerous since the increase in braking times were minimal. Limitations of this study include the important fact that driving simulation is not real-time driving. In order to assess the validity of the driving simulator used in this study, a similar experimental study during real-time driving was thus devised.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects between 25 to 60 years old
* Possession of a valid Quebec driver's license
* Driving for at least 5 years
* Exclusively use the right foot for accelerating and braking

Exclusion Criteria:

* Visual acuity deficits or other visual problems uncompensated
* History of drug or alcohol abuse
* Use of psychotropic drugs
* Any illness of the central nervous system such as epilepsy
* Sleep disorders
* Metabolic problems
* Cardiovascular disease
* Cerebrovascular disease
* Peripheral vascular disease
* Psychiatric illness
* Renal disease
* Musculoskeletal disease
* Motion sickness

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Braking performances during real-time driving. | Two years.
  The braking performances are assessed using (1) the median foot movement time, (2) the median brake reaction time and (3) the median total braking time.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Cabana, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (2):
- Canada (2):
  - Centre de recherche sur le vieillissement, Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec